CLINICAL TRIAL: NCT05903105
Title: The Preference of a Culturally and Linguistic Diverse (CALD) Population for Second Line OAB Therapy: a Discrete Choice Experiment
Brief Title: Diversity in Patients With OAB
Acronym: DOAB
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Sint-Lucas Gent (Other); AZ Jan Palfijn Gent (Other); Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0337
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder; Diversity; Onabotulinum Toxin A; Sacral Neuromodulation; Discrete Choice Experiment
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overactive Bladder: Adult patients with overactive bladder
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients fill in a questionnaire

SUMMARY:
An overactive bladder (OAB) is a condition characterized by frequent en nightly voiding, small bladder capacity and the occurrence of sudden urge to void, with or without urinary incontinence. The prevalence of OAB with bothersome complaints is around 11% in women and 9% in men with an increasing incidence with age. OAB is not an illness or disease but nevertheless had a significant impact on both the individual as society. First-line treatment for OAB consists out of behavioral and physiotherapy. Anticholinergic medication can be associated to improve bothersome symptoms, but has the downside of causing unwanted side effects. If the formentioned treatment is not sufficient, second line treatment can be discussed. Depending on the patient's characteristics and the physician's preference intravesical injections of Botox or the implantation of a sacral neuromodulator (SNM) can be considered.

Both options are equal and effective, but many individual differences exist in preference. Regarding outcome, some factors have been described to prefer one therapy above the other, for example in case of concomitant fecal incontinence, frequent urinary tract infections,… The personal preference of doctors and patients has been investigated, but currently no study has focused on therapy preference in a culturally and linguistic divers (CALD) population. The latter broadly describes a population with ethnical, cultural, religious and/or language characteristics and is a general accepted measure of diversity.

In the current study, the investigators aim to describe the different (dis)advantages of both second line treatments for OAB in a discrete choice experiment. The study population will consist of a diverse group of patients with OAB from different hospitals. The goal is to investigate if CALD patients make a different choice in treatment and what factors contribute to that decision in order to provide more tailored information regarding the treatment options in the future. Taking a patient's context into account in the shared decision making between a patient and physician increases therapy compliance and satisfaction of the chosen treatment.

The total questionnaire will consist out of general demographic info, the EQ-5D, the International Consultation on Incontinence Questionnaire (ICIQ)-OAB and the discrete choice questionnaire in which patients make a choice between two fictional treatment options consisting of a combination of different therapy characteristics. The questionnaire will be translated into different languages in order to lower the threshold for participation.

ELIGIBILITY:
Inclusion Criteria:

* OAB
* Adult

Exclusion Criteria:

* SNM or Botox in history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with an overactive bladder are eligible to participate in the study. Patients who received intravesical botox or had/have a SNM implanted are not eligible.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Discrete choice questionnaire | 1 hour
  Patients choose between two fictive therapies, each option comes with it's own botox and sacral neurmodulator (SNM) characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East-Fanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided